CLINICAL TRIAL: NCT03321240
Title: Study of Predictive Biomarkers for Rational Management of Drug-resistant Epilepsy Associated With Focal Cortical Dysplasia
Acronym: SPREAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6647
Record Dates: First submitted 2017-10-16; First posted 2017-10-25 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Refractory Epilepsy; Focal Epilepsy; Focal Cortical Dysplasia
Keywords: focal cortical dysplasia; Pronostic; Epilepsy surgery; Epiletogenicity index; SEEG
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsies, Partial; Focal Cortical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample and resected brain tissue specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The SEEG group: Group with the SEEG analysis
  Interventions: Procedure: visual and quantitative SEEG signal analysis; Procedure: Resective epilepsy surgery procedure
- The direct surgery group: Group with a direct surgery
  Interventions: Procedure: Resective epilepsy surgery procedure

INTERVENTIONS:
Procedure: visual and quantitative SEEG signal analysis — signal SEEG analysis
  Groups: The SEEG group
Procedure: Resective epilepsy surgery procedure — Surgical removal of the epileptogenic brain area

SUMMARY:
Focal Cortical Dysplasias (FCDs) are neurodevelopmental disorders that represent a major cause of early onset drug-resistant epilepsies with cognitive and behavioral impairments, carrying a lifelong perspective of disability and reduced quality of life. Despite a major medical and socio-economic burden, rationale therapeutic strategies are still under debate. Surgical removal of the epileptogenic brain area (Epileptogenic Zone) is the most successful treatment, yet it fails to control FCD-associated seizures in as much as 40% of cases. Precise definition and complete resection of the Epileptogenic Zone are the main determinants of outcome. In current practice of French centers, up to 80% FCD-patients require an intracranial EEG (icEEG) recording to accurately define the epileptogenic zone. However, the indications for icEEG in MRI-visible FCD remain empirical and are essentially based on expert opinion.

ELIGIBILITY:
Inclusion Criteria:

* Adult or pediatric patient suffering from drug-resistant focal epilepsy;
* Age more than 2 years old;
* Brain MRI suggestive of FCD or normal;
* Standardized presurgical evaluation available including medical history, scalp video-EEG, 3T MRI, FDG-PET, Neuropsychological tests;
* Inpatient in one of the participating centers for recording seizure during long term scalp video-EEG and / or SEEG-monitoring;
* Resective surgery with a minimal post-operative follow-up of 12 months;
* Histopathologic evidence for FCD or non-pathologic findings (normal histology or mMCD type II).
* Patient, parents or legally representative who have given written informed consent to allow the study data collection procedures.

Exclusion Criteria:

* Brain MRI suggestive of another type of lesion;
* Difficulty to read or understand French, or inability to understand the information;
* Pregnant or breastfeeding woman;
* Subject under judicial protection.
* Other lesion discovered on histological examination;
* FCD type 3, dual pathology, ambiguous or unavailable neuropathological findings
* Lack of longitudinal pre- and post-surgical follow-up.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult or pediatric (Age more than 2 years old) patients attending tertiary epilepsy center for presurgical evaluation of refractory focal epilepsy compatible with FCD
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of seizure-free patients (Engel class I) at 12-months follow-up after resective surgery. | 12 month

SECONDARY OUTCOMES:
Proportion of each of six seizure-onset pattern types within each of three histologically defined subgroups (FCD type I, FCD type II, non-pathologic findings). | 12 month
Duration of epilepsy before surgery in patients with focal and network epileptogenic zone (defined by EI) | 12 month
Topographic distribution of structures that disclose high Epileptogenicity Index values (EI>0.4), of structures with maximal interictal HFO rates and of structures showing interictal/preictal functional connectivity alterations | 12 month

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Michallon Hospital, Grenoble
  - Hôpital Roger Salengro, Lille
  - Hospices Civils de Lyon, Lyon
  - Timone Hospital, Marseille
  - University Hospital of Nancy, Nancy
  - GH Pitie-Salpêtrière-Charles Foix, Paris
  - Necker-Enfants Malades Hospital, Paris
  - Rothschild Foundation, Paris
  - CHU Rennes, Rennes
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Pierre Paul Riquet, Toulouse